CLINICAL TRIAL: NCT02100007
Title: A Phase Ib Open Label Study of the Safety and Tolerability of ME-344 Given in Combination With Topotecan (Hycamtin®) in Patients With Solid Tumors
Brief Title: ME-344 Given in Combination With Hycamtin® in Patients With Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: lack of efficacy
Sponsor: MEI Pharma, Inc. (Industry)
Collaborators: SCRI Development Innovations, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ME-344-002
Record Dates: First submitted 2014-03-24; First posted 2014-03-31 (Estimated); Results first posted 2017-10-02 (Actual); Last update posted 2017-10-02 (Actual); Status verified 2015-08

CONDITIONS: Solid Tumors
Keywords: solid tumors; relapsed; advanced; metastatic; small cell lung cancer; ovarian cancer; refractory
MeSH Terms: conditions — Recurrence; Neoplasm Metastasis; Small Cell Lung Carcinoma; Ovarian Neoplasms | interventions — ME-344; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ME-344 (Experimental): ME-344 IV, 10 mg/kg on Days 1, 8, 15 and 22 of each 28 day cycle Topotecan IV, 4 mg/m2 on Days 1, 8 and 15 of each 28 day cycle
  Interventions: Drug: ME-344; Drug: Topotecan

INTERVENTIONS:
Drug: ME-344 — Part 1: ME-344 IV at 10 mg/kg on Days 1, 8, 15, and 22 of each 28-day cycle. Part 2: ME-344 IV at the dose defined in Part 1 on Days 1, 8, 15, and 22 of each 28 day cycle.
  Patients will be allowed to continue receiving ME-344 infusions weekly according to the assigned dose level as long as there is clinical benefit to the patient as assessed by the Investigator.
  Other Names: open label
Drug: Topotecan — Part 1: Topotecan 4 mg/m2 i.v. weekly on Days 1, 8 and 15 of each 28-day cycle. Part 2: Topotecan 4 mg/m2 i.v. weekly on Days 1, 8 and 15 of each 28-day cycle.
  Other Names: Hycamtin®

SUMMARY:
The purpose of this study is to determine the safety and tolerability of ME-344 when given in combination with Hycamtin® in patients with solid tumors

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic confirmed locally advanced or metastatic small cell lung cancer, ovarian cancer, or cervical cancer (Part 1); small cell lung cancer and ovarian cancer (Part 2)
* Patients with ovarian and small cell lung cancer must have failed initial therapy
* Patients with carcinoma of the cervix must have advanced disease not amenable to curative surgery and/or radiation therapy
* Patients may not have received more than 4 prior regimens of therapy
* Patients may not previously have received irinotecan, topotecan or other topoisomerase I inhibitor
* ECOG Performance status 0-1 (Appendix B)
* A minimum life expectancy of 12 weeks
* Adequate bone marrow, hepatic and renal function as evidenced by:

  * Absolute neutrophil count (ANC) > 1.5 x 109/L
  * Platelet count > 100 x 109/L
  * Hemoglobin > 9.0 g/dL
  * Serum bilirubin < 1.5 x ULN
  * AST/ALT (SGOT/SGPT) < 2.5 x ULN for the reference laboratory or < 5 x --ULN in the presence of liver metastases
  * Serum creatinine < 1.5 x ULN or creatinine clearance ≥ 60 mL/min as measured by institutional standards
* At least 21 days must have elapsed prior to Day 1 Cycle 1, since any radiotherapy, immunotherapy or following major surgery; any surgical incision should be completely healed. At least 14 days must have elapsed prior to Day 1 Cycle 1 since "limited palliative radiotherapy", defined as a course of therapy encompassing <25% total bone marrow volume and not exceeding 30 GY.

Exclusion Criteria:

* Patients with tumor involvement of the Central Nervous System (CNS). SCLC patients with previously treated CNS lesions must have stable CNS disease for at least 4 weeks
* Patients with uncontrolled infection or systemic disease
* Patients with clinically significant cardiac disease not well controlled with medication (e.g., congestive heart failure, symptomatic coronary artery disease e.g. angina, and cardiac arrhythmias) or myocardial infarction within the last 12 months
* Patients who have toxicity from last prior therapy that has not recovered to at least Grade 1, with the exception of Grade 2 alopecia
* Patients who have had any chemotherapy regimens, biologic, or targeted therapies within the 2 weeks prior to Cycle 1 Day 1
* Patients with any neuropathy > Grade 1
* Patients with known hypersensitivity to any components of ME-344 or topotecan study drug product
* Patients with known human immunodeficiency virus (HIV) or Hepatitis B or C (active, previously treated or both)
* Patients with a history of solid organ transplantation
* Patients with presence of concurrent or active malignant disease (other than disease under study) within the last 12 months with the exception of adequately treated in-situ carcinomas, basal or squamous cell carcinoma, or non-melanomatous skin cancer.

Patients with any psychiatric disorder or social or geographic situation that would preclude study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-04; Primary Completion 2016-01 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Ghalie, MD, Study Director — MEI Pharma, Inc.
Locations (10):
- United States (8):
  - Pinnacle Oncology Hematology, Scottsdale, Arizona
  - University of Colorado Cancer Center, Aurora, Colorado
  - Northwestern University, Chicago, Illinois
  - Oncology Hematology Care, Cincinnati, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Medical University of South Carolina, Charleston, South Carolina
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - University of WA Seattle Cancer Care Alliance, Seattle, Washington
- United Kingdom (2):
  - The Bays St Mary's Hospital, London, England
  - Sarah Cannon Research Instititute UK, London, England

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor website — http://www.meipharma.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was open to recruitment from April 30, 2014 through December 7, 2015 at 7 investigational sites in the USA and 2 sites in the United Kingdom. Forty-six patients were enrolled. The study was conducted in two parts. Fourteen (14) patients enrolled in Part 1 and 32 subjects were enrolled in Part 2.
Pre-assignment Details: Fifty-eight (58) potential participants were screened; 46 subjects passed screening and were enrolled in the study.
Groups:
- ME-344: ME-344 IV, 10 mg/kg on Days 1, 8, 15 and 22 of each 28 day cycle Topotecan IV, 4 mg/m2 on Days 1, 8 and 15 of each 28 day cycle
  ME-344: Part 1: ME-344 IV at 10 mg/kg on Days 1, 8, 15, and 22 of each 28-day cycle.
  Part 2: ME-344 IV at the dose defined in Part 1 on Days 1, 8, 15, and 22 of each 28 day cycle.
  Patients will be allowed to continue receiving ME-344 infusions weekly according to the assigned dose level as long as there is clinical benefit to the patient as assessed by the Investigator.
  Topotecan: Part 1: Topotecan 4 mg/m2 i.v. weekly on Days 1, 8 and 15 of each 28-day cycle.
  Part 2: Topotecan 4 mg/m2 i.v. weekly on Days 1, 8 and 15 of each 28-day cycle.
Period: Overall Study
Arm/Group | ME-344
Started | 46
Completed | 46
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The study was conducted in two parts. Fourteen (14) patients enrolled in Part 1 and 32 subjects were enrolled in Part 2.
Arm/Group | ME-344
Number analyzed (Participants) | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 34
  >=65 years | 12
Age, Continuous [Median (Full Range); unit: Years] | 59.5 [26 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 41
  Unknown or Not Reported | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 42
  Black or African American | 1
  Asian | 2
  Other | 1
Region of Enrollment [Number; unit: participants]
  United States | 38
  United Kingdom | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events
Description: The AE Profile will be determined by the number of AEs regardless of severity
Time Frame: Through study completion- an average of 2 years
Population: 46 subjects received > 2 doses of ME-344 and topotecan and were eligible for DLT analysis.
Measure: Number; unit: adverse events
Arm/Group | ME-344
Number analyzed (Participants) | 46
adverse events | 595

2. Primary Outcome: Number of Serious Adverse Events
Description: The SAE Profile will be determined by the number of SAEs
Time Frame: Through study completion- an average of 2 years
Population: 46 subjects received > 2 doses of ME-344 and topotecan and were eligible for DLT analysis.
Measure: Number; unit: SAEs
Groups:
- ME-344: ME-344 IV, 10 mg/kg on Days 1, 8, 15 and 22 of each 28 day cycle ...
Arm/Group | ME-344
Number analyzed (Participants) | 46
SAEs | 23

3. Secondary Outcome: Maximum Plasma Concentration (Cmax)
Description: Peak Plasma Concentration (Cmax) of ME-344 in combination with topotecan
Time Frame: Cycle 1 Day 1, at 0, .5, 1, 2, 4, 6 and 24 hours post-dose and Day 15 at 0 and end of infusion
Population: Pharmacokinetic parameters for ME-344 in plasma were calculated based on the plasma concentration data from 13 patients who received treatment in Part 1 of the study.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ME-344
Number analyzed (Participants) | 12
ng/mL | 20880 (8201.3)

4. Secondary Outcome: Time to Maximum Plasma Concentration for ME-344 (Tmax)
Description: Various pharmacokinetic parameters for ME-344 in plasma were calculated based on the plasma concentration data.
Time Frame: Cycle 1 Day 1, at 0, .5, 1, 2, 4, 6 and 24 hours post-dose and Day 15 at 0 and end of infusion
Population: Samples were collected from patients in Part 1 of the study for measurement of plasma concentration of ME-344. Samples were collected from 13 patients in Part 1
Measure: Mean (Full Range); unit: hours
Arm/Group | ME-344
Number analyzed (Participants) | 13
hours | 0.5 [0.48 to 2.02]

5. Secondary Outcome: Minimum Plasma Concentration (Cmin) of ME-344
Description: Various pharmacokinetic parameters for ME-344 in plasma were calculated based on the plasma concentration data.
Time Frame: Cycle 1 Day 1, at 0, .5, 1, 2, 4, 6 and 24 hours post-dose and Day 15 at 0 and end of infusion
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ME-344
Number analyzed (Participants) | 13
ng/mL | 25.3 (12.824)

6. Secondary Outcome: Mean Terminal Half-life (t 1/2)
Description: Various pharmacokinetic parameters for ME-344 in plasma were calculated based on the plasma concentration data.
Time Frame: Cycle 1 Day 1, at 0, .5, 1, 2, 4, 6 and 24 hours post-dose and Day 15 at 0 and end of infusion
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | ME-344
Number analyzed (Participants) | 13
hours | 5.301 (2.0114)

7. Secondary Outcome: Estimate Overall Response Rate for ME-344 Given in Combination With Topotecan
Description: Overall response rate was defined as the total number of patients with Complete Response plus Partial Response. All efficacy assessments were to include a baseline assessment and follow-up assessments at a minimum of every 8 weeks for the first 6 cycles, then every 12 weeks thereafter, while receiving study drug. Tumor response and progression-free survival were assessed using RECIST 1.1 criteria or GCIG criteria for CA-125 levels.
Time Frame: Response was assessed throughout the trial up to 13 months
Population: Part 1 (N =12), Part 2 (N=29)
Measure: Number; unit: participants
Arm/Group | ME-344
Number analyzed (Participants) | 41
participants | 1

8. Secondary Outcome: Estimate the Overall Survival (OS)
Description: 41 subjects were analysed. Overall survival is defined as the first day of study drug administration to death.
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ME-344
Number analyzed (Participants) | 41
months | 3.7 [2.8 to 5.4]

ADVERSE EVENTS:
Time Frame: The occurrence of adverse events was assessed throughout the trial, up to 13 months.
Description: Forty-six patients were enrolled in the trial and were to receive both ME-344 and topotecan. Forty-five subjects received both drugs, 1 subject received only ME-344
Arm/Group | ME-344
All-Cause Mortality (participants affected / at risk) | 6/46
Serious Adverse Events (participants affected / at risk) | 17/46
Other Adverse Events (participants affected / at risk) | 46/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ME-344 (N=46)
Procedural Pain (Injury, poisoning and procedural complications) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Fatique (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1)
Bacteremia (Infections and infestations) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 1 (2)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (3)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ME-344 (N=46)
Hypertension (Vascular disorders) | 19 (27)
Fatigue (General disorders) | 30 (42)
Asthenia (General disorders) | 7 (11)
Chest pain (General disorders) | 6 (10)
Chest discomfort (General disorders) | 5 (7)
Muscosal inflammation (General disorders) | 3 (5)
Oedema peripheral (General disorders) | 3 (3)
Peripheral swelling (General disorders) | 3 (3)
Pyrexia (General disorders) | 3 (4)
Anxiety (Psychiatric disorders) | 3 (3)
Infusion related reaction (Injury, poisoning and procedural complications) | 4 (6)
Weight decreased (Investigations) | 9 (12)
White blood cell count decreased (Investigations) | 6 (13)
Neutrophil count decreased (Investigations) | 5 (11)
Platelet count decreased (Investigations) | 5 (25)
QTc Prolonged (Investigations) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 21 (45)
Thrombocytopenia (Blood and lymphatic system disorders) | 18 (33)
Anaemia (Blood and lymphatic system disorders) | 16 (31)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Headache (Nervous system disorders) | 6 (6)
Dizziness (Nervous system disorders) | 5 (5)
Paraesthesia (Nervous system disorders) | 4 (5)
Nausea (Gastrointestinal disorders) | 22 (34)
Diarrhoea (Gastrointestinal disorders) | 21 (25)
Vomiting (Gastrointestinal disorders) | 18 (29)
Constipation (Gastrointestinal disorders) | 15 (19)
Abdominal pain (Gastrointestinal disorders) | 7 (12)
Abdominal pain lower (Gastrointestinal disorders) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3)
Dysuria (Renal and urinary disorders) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 (6)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 19 (20)
Hypokalemia (Metabolism and nutrition disorders) | 6 (24)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (4)
Hyponatremia (Metabolism and nutrition disorders) | 3 (5)
Urinary tract infection (Infections and infestations) | 5 (5)
Upper Respiratory Tract Infection (Infections and infestations) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Each PI has a CDA in place that restricts them from discussing the results of the clinical study at a scientific meeting or any other public or private forum or to publish in a scientific or academic journal the results of the clinical study without the approval of the Sponsor Company (MEI Pharma Inc.).